CLINICAL TRIAL: NCT06818981
Title: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial of Post-Operative Steroids After Sleep Surgery
Brief Title: Post-Operative Steroids After Sleep Surgery
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Mohamed Abdelwahab, Assistant Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Pro00138969
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: Pain; Sleep Disorders; Surgery
MeSH Terms: conditions — Sleep Apnea, Obstructive; Pain; Sleep Wake Disorders | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- 3 doses of intravenous 8mg dexamethasone with 3 doses of oral 8mg dexamethasone (Experimental): Experimental drug administered both intravenously and orally
  Interventions: Drug: 8mg dexamethasone
- 3 doses of intravenous 8mg dexamethasone with 3 doses of placebo (Other): Experimental drug administered intravenously, while the placebo is administered orally
  Interventions: Drug: 8mg dexamethasone
- 3 doses of intravenous placebo with 3 doses of oral 8mg dexamethasone (Other): Placebo administered intravenously, while the experimental drug is administered orally
  Interventions: Drug: 8mg dexamethasone
- 3 doses of intravenous placebo with 3 doses of placebo (Placebo Comparator): Placebo administered both intravenously and orally
  Interventions: Drug: 8mg dexamethasone

INTERVENTIONS:
Drug: 8mg dexamethasone — Minimal research exists on how to treat pain, odynophagia, and dysphagia in sleep surgery patients. One study by Williams et al. evaluated the use of a one-time dose of intravenous or intramuscular dose of steroids versus placebo after uvulopalatopharyngoplasty but did not find a clinically significant difference between the two groups postoperatively. However this study mentioned that their current intervention was too short and that a longer-term steroid intervention could be beneficial. This is the goal of this intervention.
  Other Names: Decadron

SUMMARY:
The primary objective of this randomized, placebo-controlled, double-blind study will be to determine if postoperative steroids significantly improve subjects' pain compared to a placebo after undergoing sleep surgery. The secondary objective is to determine if this same course of steroids improves how quickly subjects can tolerate a regular diet after surgery. Further, another secondary objective is to see if this will decrease a patient's postoperative narcotic usage. Investigators also will assess sleepiness, nasal breathing, and eustachian tube dysfunction (ETD) after the procedure using the validated measures Preoperative Epworth Sleepiness Scale (ESS), Nasal Obstruction Symptom Evaluation Survey (NOSE), and Eustachian Tube Dysfunction Questionnaire (ETDQ-7) with an objective to see if these improve more or quicker in patients who receive postoperative steroids. Investigators hypothesize that postoperative steroids will significantly decrease a patient's pain quicker in their recovery, allow them to tolerate more oral intake early in their recovery, allow them to tolerate a regular diet earlier in their recovery, and reduce their postoperative narcotic usage. Investigators hypothesize that postoperative steroids will also improve patients' ESS, NOSE, and ETD scores postoperatively, but Investigators do not believe postoperative steroids will affect the oropharyngeal bleeding rate of patients. This study will provide pilot data to determine if postoperative steroids and what dosage should be part of a standardized postoperative regimen in patients undergoing sleep surgery.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a multifactorial disease that negatively affects almost every system in the body. While continuous positive airway pressure (CPAP) can be used as an effective treatment, there are many reasons that patients cannot tolerate CPAP, including claustrophobia, rhinitis sicca, ineffectiveness, and manufacturer recalls that most recently have even been fatal. Therefore, sleep surgery continues to be an increasingly utilized treatment option for patients with OSA who cannot tolerate or obtain CPAP. However postoperatively, patients typically complain of significant pain, sometimes requiring a significant course of narcotic pain medication, odynophagia, and dysphagia. These side effects often can make patients hesitant to pursue sleep surgery and carry the risk of patients becoming dehydrated and malnourished postoperatively, which can lead to representation to the Emergency Department. Minimal research currently exists on how to improve treating pain, odynophagia, and dysphagia in this patient population. One study by Williams et al. evaluated the use of a one-time dose of intravenous or intramuscular dose of steroids versus placebo after uvulopalatopharyngoplasty but did not find a clinically significant difference between the two groups postoperatively. However, in their study, they mention that likely their intervention was too short, and that further investigation into a longer course of steroid treatment, our current intervention for this study, could potentially show clinically significant improvements. Furthermore, there have been a few randomized controlled trials showing that a course of steroids improve pain and narcotic consumption after tonsillectomy in adults. However, no research has studies the postoperative effects of steroids on other sleep surgeries, such as palatopharyngoplasty, hypoglossal nerve stimulation, genioglossus advancement, or maxillomandibular advancement. Investigators hypothesize that postoperative steroids will be superior to no steroids in terms of pain, dysphagia, and narcotic usage.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older
* Undergoing sleep surgery, specifically palatopharyngoplasty, tonsillectomy with or without adenoidectomy, uvulectomy, hypoglossal nerve stimulation, genioglossal advancement, or maxillomandibular advancement
* Ability to complete all study questions in English

Exclusion Criteria:

* Any self-reported allergies to corticosteroids
* Intra-operative surgical or anesthetic complication
* Pre-operative steroid use (defined as any steroid use greater than three days duration within 30 days prior to sleep surgery)
* Inability to perform study due to underlying medical condition
* Inability to answer postoperative questionnaires due to underlying medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain control | 2 weeks
  As determined by a validated visual analog scale, with scores being scaled from 0 to 10, with 0 being the lowest score (no pain) and 10 being the highest score (most extreme amount of pain)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Poupore, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lachance M, Lacroix Y, Audet N, Savard P, Thuot F. The use of dexamethasone to reduce pain after tonsillectomy in adults: a double-blind prospective randomized trial. Laryngoscope. 2008 Feb;118(2):232-6. doi: 10.1097/MLG.0b013e318159a5cc. PMID 18043492
- [Background] Stewart R, Bill R, Ullah R, McConaghy P, Hall SJ. Dexamethasone reduces pain after tonsillectomy in adults. Clin Otolaryngol Allied Sci. 2002 Oct;27(5):321-6. doi: 10.1046/j.1365-2273.2002.00588.x. PMID 12383289
- [Background] Williams PM, Strome M, Eliachar I, Lavertu P, Wood BG, Vito KJ. Impact of steroids on recovery after uvulopalatopharyngoplasty. Laryngoscope. 1999 Dec;109(12):1941-6. doi: 10.1097/00005537-199912000-00008. PMID 10591351
- [Background] Abdelwahab M, Marques S, Howard J, Huang A, Lechner M, Olds C, Capasso R. Incidence and risk factors of chronic opioid use after sleep apnea surgery. J Clin Sleep Med. 2022 Jul 1;18(7):1805-1813. doi: 10.5664/jcsm.9978. PMID 35393936
- [Background] Shah RR, Thaler ER. Base of Tongue Surgery for Obstructive Sleep Apnea in the Era of Neurostimulation. Otolaryngol Clin North Am. 2020 Jun;53(3):431-443. doi: 10.1016/j.otc.2020.02.006. Epub 2020 Apr 23. PMID 32334869
- [Background] Barrera JE. Skeletal Surgery for Obstructive Sleep Apnea. Sleep Med Clin. 2018 Dec;13(4):549-558. doi: 10.1016/j.jsmc.2018.07.006. PMID 30396448
- [Background] Smith DF, Cohen AP, Ishman SL. Surgical management of OSA in adults. Chest. 2015 Jun;147(6):1681-1690. doi: 10.1378/chest.14-2078. PMID 26033129
- [Background] Kapur VK, Auckley DH, Chowdhuri S, Kuhlmann DC, Mehra R, Ramar K, Harrod CG. Clinical Practice Guideline for Diagnostic Testing for Adult Obstructive Sleep Apnea: An American Academy of Sleep Medicine Clinical Practice Guideline. J Clin Sleep Med. 2017 Mar 15;13(3):479-504. doi: 10.5664/jcsm.6506. PMID 28162150